CLINICAL TRIAL: NCT00157131
Title: A Study To Evaluate the Safety and Efficacy of Fibrin Sealant With 4IU/mL Thrombin, Vapor Heated, Solvent Detergent Treated (FS 4IU VH S/D) to Adhere Tissues and Improve Wound Healing
Brief Title: Safety and Efficacy Study of FS 4 IU VH S/D (Fibrin Sealant With 4IU/mL Thrombin, Vapor Heated, Solvent/Detergent Treated) to Adhere Split Thickness Skin Grafts and Improve Wound Healing in Burn Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Baxter Healthcare Corporation (Industry)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 550201
Record Dates: First submitted 2005-09-08; First posted 2005-09-12 (Estimated); Last update posted 2017-04-20 (Actual); Status verified 2017-04

CONDITIONS: Deep Partial or Full Thickness Wounds
Keywords: autologous sheet skin grafts; FS 4IU VH S/D; skin grafts; burn
MeSH Terms: conditions — Burns | interventions — Fibrin Tissue Adhesive; Sutures

STUDY DESIGN:
Who Masked: Outcomes Assessor

ARMS (2):
- FS 4IU VH S/D (Experimental): FS 4IU VH S/D was administered intraoperatively to the wound bed by spray application using the TISSOMAT and Spray Set. Only the DUPLOJECTvii system and Spray Set (connection tube with sterile filter and spray head) device was used for simultaneous spray application of the study product. A thin layer of FS 4IU VH S/D was applied to the wound bed using a "painting motion" from side to side to achieve coverage. The recommended dosing volume was 2.0 to 4.0 mL/100 cm2. One 2-mL pack (4 mL total volume) of FS 4IU VH S/D applied using the TISSOMAT and Spray Set was sufficient to coat a wound bed of 100-200 cm2.
  Interventions: Biological: Fibrin Sealant, ARTISS 4IU/ml VH SD
- Staples (Active Comparator): Staples are the current standard of care in burn surgery and are well accepted as the control in this type of study.
  Interventions: Other: Staples

INTERVENTIONS:
Biological: Fibrin Sealant, ARTISS 4IU/ml VH SD — FS 4IU VH S/D, a two-component fibrin sealant with 4 IU/mL human thrombin, vapor heated, solvent detergent treated, provided in a frozen, ready-to-use formulation. Administration by a topical spray application using the TISSOMAT device and Spray Set.
  Arms: FS 4IU VH S/D
Other: Staples — Administration by mechanical/multiple point fixation.
  Arms: Staples

SUMMARY:
The primary objective of this study is to evaluate skin graft adherence and wound healing in burn patients to evaluate whether FS 4IU VH S/D is equivalent or superior to the current standard of care (staples). The primary endpoint is achievement of complete (100%) wound closure within 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or their legal representatives, who have read, understood and signed a written informed consent.
* Subjects of either sex.
* Female subjects of childbearing potential with a negative urine or serum pregnancy test on admission.
* Subjects who are <= 65 years of age including pediatric subjects of all ages.
* Subjects with total burn wounds measuring <= 40% TBSA.
* Subjects with a contiguous deep partial thickness/full thickness wound, between 2% and 8% TBSA or two comparable, bilateral wounds each measuring between 1% and 4% TBSA.
* Wounds designated as test sites require autologous sheet skin grafts with a thickness of 8/1000" - 16/1000"
* Subjects who are able, and willing to comply with the procedures required by the protocol.

Exclusion Criteria:

* Subjects with electrical burns.
* Subjects with chemical burns
* Digits and genitalia are excluded as test sites.
* Subjects with infection at test area/test sites.
* Subjects with test sites previously randomized and treated in this study.
* Subjects with venous or arterial vascular disorder that directly affects a designated test area/test site.
* Subjects with pre-existing hemolytic anemia
* Subjects with diabetes mellitus.
* Subjects with documented history of pathologically or pharmacologically induced immune deficiency.
* Subjects judged to be chronically malnourished.
* Subjects that are judged to have significant pulmonary compromise.
* Subjects receiving systemic corticosteroids within 30 days prior to skin grafting (not including inhaled steroids).
* Subjects with known or suspected hypersensitivity to bovine proteins.
* Subjects participating in another clinical trial that is evaluating an unapproved drug or device.

Max Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 150 (Actual)
Dates: Start 2004-06; Primary Completion 2007-02 (Actual); Study Completion 2007-02 (Actual)

PRIMARY OUTCOMES:
Complete wound closure by Day 28 after treatment with either FS 4IU VH S/D or staples as determined by a blinded independent review of the Day 28 photographs | 28 days after treatment
Adverse experiences (AEs) deemed possibly or probably related to treatment with FS 4IU VH S/D | 12 months after treatment

SECONDARY OUTCOMES:
Presence of hematoma/seroma on Day 1 | 1 day after treatment
Percent area of hematoma/seroma on Day 1 | 1 day after treatment
100% engraftment by Day 5 | 5 days after treatment
Percent area of engraftment on Day 5 | 5 days after treatment
Complete wound closure by Day 14 | 14 days after treatment
Percent area of closure by Days 14 and 28 | 14 and 28 days after treatment
Scar maturation assessed by blinded Vancouver Scar Scale evaluations on Months 3, 6, 9, and 12 | 3, 6, 9, and 12 months after treatment

CONTACTS AND LOCATIONS:
Overall Officials: David Greenhalgh, MD, Principal Investigator — Shriners Hospitals for Children, Northern Calif.
Locations (17):
- United States (17):
  - Birmingham, Alabama
  - Mobile, Alabama
  - Phoenix, Arizona
  - Orange, California
  - Sacramento, California
  - San Diego, California
  - Gainesville, Florida
  - Maywood, Illinois
  - Springfield, Illinois
  - Baltimore, Maryland
  - Lincoln, Nebraska
  - Cincinnati, Ohio
  - Allentown, Pennsylvania
  - Philadelphia, Pennsylvania
  - Lubbock, Texas
  - Seattle, Washington
  - Madison, Wisconsin

REFERENCES:
- [Result] Foster K, Greenhalgh D, Gamelli RL, Mozingo D, Gibran N, Neumeister M, Abrams SZ, Hantak E, Grubbs L, Ploder B, Schofield N, Riina LH; FS 4IU VH S/D Clinical Study Group. Efficacy and safety of a fibrin sealant for adherence of autologous skin grafts to burn wounds: results of a phase 3 clinical study. J Burn Care Res. 2008 Mar-Apr;29(2):293-303. doi: 10.1097/BCR.0b013e31816673f8. PMID 18354285